CLINICAL TRIAL: NCT05897983
Title: Efficacy of Transcutaneous Electrical Nerve Stimulation Plus Rocabado Exercises on Temporomandibular Joint Dysfunction After Head and Neck Surgeries
Brief Title: Tens and Rocabado Exercises on TMJ Dysfunction
Acronym: TMJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Mohamed Mohamed Elattar, master, Assistant lecturer of physical therapy., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 782015
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rocabado exercises plus TENS (Experimental): Rocabado exercises plus TENS and traditional exercises For 8 weeks,Rocabado exercises form of 2 parts , 6×6×6 exercises part are repeated 6 times a day for 20 minutes for each repetition and mobilization exercises are done by the therapist 3 times a week for 20 min ,each mobilization is performed for 10-15 times and repeated for 5-6 times. TENS is used, with a maximum frequency of 120 Hz and an intensity range of 0 to 99.5 mA and the pulse width is between 50-200 microseconds, The TENS will be applied for 20 min 2 sessions/week for 8 weeks, Traditional exercises are passive , active Rom exercises and massage, these exercises are performed for 30 minutes and repeated 2 times daily
  Interventions: Other: Rocabado exercises plus TENS device
- Rocabado exercises (Experimental): Rocabado exercises part (1): 6×6×6 exercises are (1).The rest position of the tongue , (2). Shoulder retraction exercises, (3). Stabilized head flexion ,( 4). The axial extension of the neck , (5).Control of TMJ rotation , (6).Rhythmic stabilization technique . part (2): Joint mobilization) includes Distraction given with anterior glide, with anterior and lateral glide right/left & Lateral glide without distraction. Plus Traditional exercises.
  Interventions: Other: Rocabado exercises plus TENS device
- Transcutaneous electrical nerve stimulation device (Experimental): TENS is used, frequency of 120 Hz and an intensity range of 0 to 99.5 mA and the pulse width is between 50-200 microseconds. TENS electrodes are placed bilaterally on mandibular elevator muscles, on the superficial masseter muscle above the gonial angle, and bilaterally on the upper back ,The TENS will be applied for 20 min 2 sessions/week for 8 weeks. Plus Traditional exercises.
  Interventions: Other: Rocabado exercises plus TENS device

INTERVENTIONS:
Other: Rocabado exercises plus TENS device — Rocabado exercises form of 2 parts , 6×6×6 exercises part are repeated 6 times a day for 20 minutes for each repetition and mobilization exercises exercises is done by the therapist 3 times a week for 20 min ,each mobilization is performed for 10-15 times and repeated for 5-6 times. TENS is used, with a maximum frequency of 120 Hz and an intensity range of 0 to 99.5 mA and the pulse width is between 50-200 microseconds, The TENS will be applied for 20 min 3 sessions/week for 8 weeks, Traditional exercises are passive , active Rom exercises and massage, these exercises are performed for 30 minutes and repeated 2 times daily

SUMMARY:
72 patients who suffers from limited mouth opening and pain in the temporomandibular joint will be selected from oncology department in Zagazig and Cairo university hospitals: patients will be assigned randomly into three groups equal in number, 24 in each group: (group A) will receive Rocabado exercises plus transcutaneous electrical nerve stimulation and traditional exercises .(group B) will receive Rocabado exercises and traditional exercises.(groub C) will receive transcutaneous electrical nerve stimulation and traditional exercises.

DETAILED DESCRIPTION:
Patients at group A: patients will receive Rocabado exercises plus transcutaneous electrical nerve stimulation and traditional exercises For 8 weeks : Rocabado exercises form of 2 parts , 6×6×6 exercises and mobilization exercises part (1): 6×6×6 exercises are (1).The rest position of the tongue , (2). Shoulder retraction exercises, (3). Stabilized head flexion ,( 4). The axial extension of the neck , (5).Control of TMJ rotation , (6).Rhythmic stabilization technique .these 6 exercises are repeated 6 times a day for 20 minutes for each repetition.

part (2): Joint mobilization (non-thrust manipulation) includes Distraction, Distraction given with anterior glide, Distraction given with anterior and lateral glide right/left & Lateral glide without distraction. . These mobilization exercises is done by the therapist 3 times a week for 20 min ,each mobilization is performed for 10-15 times and repeated for 5-6 times.

Transcutaneous electrical nerve stimulation device(TENS):

TENS is used, with a maximum frequency of 120 Hz and an intensity range of 0 to 99.5 mA and the pulse width is between 50-200 microseconds.

TENS electrodes (diameter 35-52 mm) are placed bilaterally on mandibular elevator muscles, on the superficial masseter muscle above the gonial angle, and bilaterally on the upper back (Cacho et al.,2022).

The TENS will be applied for 20 min 2 sessions/week for 8 weeks.

Traditional exercises are passive , active Rom exercises and massage, these exercises are performed for 30 minutes and repeated 2 times daily.

1. Passive ROM exercises are done by stacked tongue depressors and number of tongue depressors are increased when improvement occur .
2. Active Rom exercises are mouth opening and closing ,side way movement and protrusion repeated for 10-15 times with holding for 5 seconds for each position.
3. Massaging for cheeks muscles for 2minutes .

Patients at group B: patients will receive Rocabado exercises and traditional exercises For 8 weeks : Rocabado exercises form of 2 parts , 6×6×6 exercises and mobilization exercises part (1): 6×6×6 exercises are (1).The rest position of the tongue ,(2). Shoulder retraction exercises, (3) .Stabilized head flexion , (4).The axial extension of the neck , (5).Control of TMJ rotation ,( 6).Rhythmic stabilization technique .these 6 exercises are repeated 6 times a day for 20 min for each repetition.

part(2): Joint mobilization (non-thrust manipulation) includes Distraction, Distraction given with anterior glide, Distraction given with anterior and lateral glide right/left & Lateral glide without distraction. . These mobilization exercises is done by the therapist 3 times a week for 20 min ,each mobilization is performed for 10-15 times and repeated for 5-6 times.

Traditional exercises are passive , active Rom exercises and massage, these exercises are performed for 30 minutes and repeated 2 times daily.

1. Passive ROM exercises are done by stacked tongue depressors and number of tongue depressors are increased when improvement occur .
2. Active Rom exercises are mouth opening and closing ,side way movement and protrusion repeated for 10-15 times with holding for 5 seconds for each position.
3. Massaging for cheeks for 2minutes .

patients at group C: patient will receive Transcutaneous electrical nerve stimulation device(TENS) and traditional exercises: TENS is used, with a maximum frequency of 120 Hz and an intensity range of 0 to 99.5 mA and the pulse width is between 50-200 microseconds.

TENS electrodes (diameter 35-52 mm) are placed bilaterally on mandibular elevator muscles, on the superficial masseter muscle above the gonial angle, and bilaterally on the upper back (Cacho et al.,2022).

The TENS will be applied for 20 min 2 sessions/week for 8 weeks.

Traditional exercises are passive , active Rom exercises and massage, these exercises are performed for 30 minutes and repeated 2 times daily.

1. Passive ROM exercises are done by stacked tongue depressors and number of tongue depressors are increased when improvement occur .
2. Active Rom exercises are mouth opening and closing ,side way movement and protrusion repeated for 10-15 times with holding for 5 seconds for each position.
3. Massaging for cheeks for 2 minutes .

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:
* Age range between 40-60 years.
* Male and female patients will participate in the study.
* All patients undergo head and neck cancer surgeries (oral cancer surgeries).
* All patients will start treatment within 6 months of radiotherapy termination.
* All patients have pain in different degrees.
* Restricted range of mouth opening < 35 mm.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Other morbid conditions in the temporomandibular region as rheumatic diseases and neurological diseases.
* Presence of other disorders involving the TMJ (e.g., myalgia, degenerative joint disease, or collagen vascular disease).
* Arthritis.
* Fracture around Temporomandibular Joint (TMJ).
* Dislocation or subluxation of TMJ.
* Inflammatory disorders of TMJ.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
. Vernier caliper: | 8 weeks
  The vernier, dial, and digital calipers give a direct reading of the distance measured with high accuracy . Vernier calipers commonly used in industry provide a precision to 0.01 mm (10 micrometres), or one thousandth of an inch. They are available in sizes that can measure up to 1,829 mm (72 in) (Agrawal et al., 2015).
Mandibular Function Impairment Questionnaire: | 8 weeks
  The Mandibular Function Impairment Questionnaire is used to assess the limitation of oral function due to mandibular function impairment. Subjects will compelete this self-reported questionnaire that comprise 17 items encompassing the difficulty of chewing hard and soft foods, taking large bites, laughing, eating certain foods, engaging in social activity, and speaking. The items are scored on a 5-point Likert scale (0-4). The overall score is calculated by dividing the sum of the item scores by 68, with a possible range of 0 to 1. A higher score denotes a more serious functional impairment. An overall score of ≤0.3 denotes a low degree, 0.3 ≤ 0.6 denotes a moderate degree, and >0.6 denotes a high degree of functional impairment( Stegenga et al.,1993).

SECONDARY OUTCOMES:
Visual Analogue Scale: | 8 weeks
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points, zero mean no pain and 10 mean sever pain (Reips and Funke,2008).

CONTACTS AND LOCATIONS:
Overall Officials: rana elattar, master, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt